CLINICAL TRIAL: NCT07042061
Title: Out-of-Hospital Cardiac Arrest Care Through Empowered and Equipped Community First Responders: Mobile External Defibrillation Investigation for Cardiac Arrest in Singapore (MEDICS).
Brief Title: Trial of Mobile External Defibrillator for Out-of-hospital Cardiac Arrest in Singapore.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Singapore Civil Defence Force (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ECOS 2024-3485
Record Dates: First submitted 2025-06-04; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Out-of-hospital Cardiac Arrest (OHCA)
Keywords: Out-of-hospital; Cardiac arrest; Automated external defibrillator; AED; Community volunteers
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AED arm (Experimental)
  Interventions: Device: Mobile external automated defibrillator

INTERVENTIONS:
Device: Mobile external automated defibrillator — A single-use, hand-held, chocolate bar sized portable AED

SUMMARY:
The goal of this clinical trial is to learn the feasibility of equipping the volunteer community responders (VCR) with the mobile external automated defibrillators (mAEDs) for the management of adults experiencing out-of-hospital cardiac arrest (OHCA) patients. It will also provide early signals if this enhanced system can help increase the frequency of defibrillation and doing it earlier. The main questions it aims to answer are:

* Can equipped VCRs apply mAEDs more frequently and earlier to potentially get more patients successfully resuscitated?
* Is this system enhancement is feasible in the long run.

Participants, the VCRs, will:

* Carry a 450 gm mAED with them all the time for up to an year and use it on an OHCA patient if and when alerted to help.
* They will hand over this single-use battery-operated device to the EMS crew for data retrieval and potential replacement
* They will be interviewed for their experience of being equipped and use of the mAED.

ELIGIBILITY:
1.1. Inclusion Criteria

Study participants must meet all the inclusion criteria to participate in this study:

1. Must be proficient in English. Able to read and understand English fluently.
2. Be aged 21-74 years of age at point of recruitment.
3. Willing and able to move rapidly to a scene that can be 400 meters away from their location.
4. Be a registered CFR with SCDF.
5. Must be active myResponder® mobile phone app user so they can receive alerts about nearby OHCA cases.

1.2. Exclusion Criteria All subjects meeting any of the following exclusion criteria will be excluded from participation in this study.

1. Not proficient in English. Cannot read and understand English.
2. Aged less than 21 and over 74 years of age.
3. Not willing to be a myResponder app user.
4. Not able to move rapidly to a scene that can be 400 meters away from their location.
5. Given the short duration of the trial, those who are pregnant will be ineligible.
6. Those experiencing any serious physical injury or handicap and those with obvious mental handicap.

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a full scale trial | Through study completion, an average of 1 year
  A validated AIM/FIM tool will be used to collect perceptions of the users and managers using a likert scale measurement reporting on feasibility and acceptability of the intervention

SECONDARY OUTCOMES:
Qualitative experiences of CFR elicited through semi-structured interviews | 1 year
  Experience of the CFRs as regards challenges faced while carrying the device and convenience when the device is needed
Qualitative experiences of CFR elicited through semi-structured interviews | 1 year
  Experience of the CFRs as regards challenges of using the new device as compared to standard of care device
Qualitative experiences of CFR elicited through semi-structured interviews | 1 year
  Responses of the patient's relatives regarding the use of the device by CFRs before and after the usage as perceived by the CFRs

OTHER OUTCOMES:
Exploratory outcome mesaures | 1 year
  Acceptability of the volunteers to carry it for 24 months (# of acceptors/# offered to carry; proportion, presented in %)
Exploratory outcome mesaures | 1 year
  Convenience to carry for an extended duration (# stopped carrying/#acceptors; proportion, presented in %)
Exploratory outcome mesaures | 1 year
  Availability when needed (# of carrying the device when needed/# acceptors; proportion, presented in %)

IPD SHARING:
Plan to Share IPD: No
The trial include government owned information and hence cannot be released.

REFERENCES:
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459